CLINICAL TRIAL: NCT00948974
Title: Variations of Cognitive Behavior Therapy for Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, James Herbert, Investigator, Drexel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18345
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2017-12

CONDITIONS: Social Anxiety Disorder
Keywords: social anxiety; treatment; Cognitive Behavioral Therapy; Acceptance and Commitment Therapy; Cognitive Therapy
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy; Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cognitive therapy (Active Comparator): cognitive therapy and exposure
  Interventions: Behavioral: Cognitive Therapy
- acceptance and committment therapy (Active Comparator): acceptance and commitment therapy and exposure
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Cognitive Therapy — Cognitive therapy (CT) highlights the identification and reappraisal of distorted or dysfunctional cognitions in the treatment of psychopathology. For example, socially anxious patients are taught to identify the thoughts and underlying beliefs that trigger strong emotional reactions (e.g., "if I attempt to initiate a conversation I'll humiliate myself"), and then replace these with more accurate, functional thoughts. There is a large body of research supporting the efficacy of CT for mood and anxiety disorders, and for social anxiety disorder in particular (Beck, 2005).
  Other Names: CT
  Arms: cognitive therapy
Behavioral: Acceptance and Commitment Therapy — ACT does not attempt to modify cognitions directly, but rather seeks to foster a mindful acceptance of whatever thoughts or feelings arise, while still pursuing specific behavioral goals. For example, the individual would be taught simply to notice the thoughts as if from a distance without attempting to modify them, and initiate a conversation. Like other newer mindfulness and acceptance-based models of CBT, ACT also expands the traditional focus on symptom reduction to include an emphasis on broader life goals. The scientific literature on ACT has expanded rapidly over the past ten years. Recent reviews conclude that it appears to be at least as effective as CT, and may work at least in part via distinct treatment mechanisms (Powers, Zum Vörde Sive Vörding, & Emmelkamp, 2009).
  Other Names: ACT
  Arms: acceptance and committment therapy

SUMMARY:
The purpose of this study is to compare the efficacy of two variants of cognitive behavioral therapy (CBT) (cognitive therapy (CT) and acceptance and commitment therapy (ACT)), for the treatment of generalized social anxiety disorder.

DETAILED DESCRIPTION:
We are recruiting a clinical sample of patients who meet diagnostic criteria (per DSM-5) for the generalized subtype of social anxiety disorder. Participants are randomly assigned to the two active intervention conditions; no placebo or sham treatments will be employed. Assessments take place at baseline, pre-treatment, mid-treatment, post-treatment, and at 3- and 12-months follow-up; participants also complete a brief weekly assessment of functioning. Treatment is administered individually by trained graduate students in clinical psychology, directly trained and supervised by the PI and Co-PI. Participants receive 12 weekly 1-hour long sessions. The study design is a 2 (treatment condition) by 5 (assessment occasion) mixed factorial design.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosable social anxiety disorder (generalized subtype per DSM-IV-TR criteria)
* aged 18-65
* working fluency in English
* residence in the greater Philadelphia area.

Exclusion Criteria:

* Pervasive developmental disability
* acute suicide potential
* inability to travel to the treatment site
* schizophrenia or other psychotic disorder
* current substance dependence
* Comorbid diagnoses of Major Depressive or other mood or anxiety disorders are acceptable ONLY if clearly secondary to the diagnosis of social anxiety disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Herbert, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Therapy | Acceptance and Committment Therapy
Started | 40 | 48
Completed | 17 | 28
Not Completed | 23 | 20
Not completed — Lost to Follow-up | 23 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Therapy | Acceptance and Committment Therapy | Total
Number analyzed (Participants) | 40 | 48 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.05 (10.25) | 29.90 (11.66) | 29.97 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 27 | 45
  Male | 22 | 21 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 10 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 22 | 21 | 43
  More than one race | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Social Phobia and Anxiety Inventory (SPAI) - Social Phobia Subscale
Description: The SPAI social phobia assess symptoms of social anxiety in the presence of (a) strangers, (b) authority figures, (c) members of the opposite sex, and (d) people in general. The subscale ranges from 32 to 192, where higher scores reflect more severe symptoms of social anxiety.
Time Frame: baseline (pre-treatment; immediately prior to beginning treatment); post-treatment (12 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Therapy | Acceptance and Committment Therapy
Number analyzed (Participants) | 17 | 28
units on a scale
  Pre-Treatment | 131.66 (19.63) | 130.17 (17.48)
  Post-Treatment | 75.47 (27.99) | 103.9 (28.72)

2. Secondary Outcome: Outcomes Questionnaire
Description: The Outcomes Questionnaire is a 45-item measure that assesses functioning and is comprised of three subscales: symptom distress, interpersonal relationships, and social role performance, that are combined to create a total score. Scores range from 45 to 180, where higher scores reflect greater levels of dysfunction.
Time Frame: baseline (pre-treatment; just before beginning treatment); post-treatment (12 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Therapy | Acceptance and Committment Therapy
Number analyzed (Participants) | 17 | 28
units on a scale
  Pre-Treatment | 120.06 (18.4) | 118.36 (25.21)
  Post-Treatment | 91.34 (24.51) | 105.54 (24.39)

3. Secondary Outcome: Behavioral Assessment Test
Description: The assessment consists of two role-played interpersonal interactions and an impromptu speech. The role-plays were video recorded for subsequent rating by two independent assessors. Using a 5-point Likert scale (1 = poor and 5 = excellent), assessors rated global social skills, which were comprised of assessments of verbal content (e.g., amount of speech during task and degree to which speech was relevant and appropriate), nonverbal skills (e.g., degree of fidgeting and eye contact; appropriateness of gestures and posture), and paralinguistic skills (e.g., appropriateness of tone, enunciation, inflection, and rate). Prior research has employed this behavioral assessment protocol (Glassman et al., 2016; Herbert et al., 2005). These results reflect global social skills, which reflect the sum of ratings of verbal, nonverbal, and paralinguistic skills. Scores range from 3 to 15 with higher scores reflecting better social skills.
Time Frame: baseline (pre-treatment; just prior to beginning treatment); post-treatment (12 weeks)
Population: A subset of randomized participants (n = 12 for ACT and n = 11 for tCBT) completed this behavioral assessment task.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Therapy | Acceptance and Committment Therapy
Number analyzed (Participants) | 11 | 12
units on a scale
  Pre-Treatment | 9.12 (2.02) | 8.33 (1.31)
  Post-Treatment | 10.2 (2.16) | 10.64 (1.37)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout each participant's 12-week participation in the study.
Description: Adverse events were monitored but no adverse events were reported by any participants.
Arm/Group | Cognitive Therapy | Acceptance and Committment Therapy
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/48
Other Adverse Events (participants affected / at risk) | 0/40 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No